CLINICAL TRIAL: NCT02445469
Title: Contribution of Magnetic Resonance Imaging (Diffusion Tensor Imaging and Magnetic Susceptibility Imaging and Resting Activation Imaging) in the Diagnosis of Parkinsonian Syndromes in Elderly Subjects.
Brief Title: Magnetic Resonance Imaging in the Diagnosis of Parkinsonian Syndromes
Acronym: PARKIMAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The results obtained are sufficient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8743
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Progressive Supranuclear Palsy; Vascular Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Parkinson's disease (Other): MRI exam of the brain
  Interventions: Other: MRI exam of the brain
- Multiple System Atrophy (Other): MRI exam of the brain
  Interventions: Other: MRI exam of the brain
- Progressive Supranuclear Palsy (Other): MRI exam of the brain
  Interventions: Other: MRI exam of the brain
- Vascular parkinsonism (Other): MRI exam of the brain
  Interventions: Other: MRI exam of the brain
- Healthy volunteers (Other): MRI exam of the brain
  Interventions: Other: MRI exam of the brain

INTERVENTIONS:
Other: MRI exam of the brain — MRI exam of the brain

SUMMARY:
Parkinsonian syndrome is clinically characterized by the presence of resting tremor, rigidity, bradykinesia and postural instability. Parkinsonian disorders include Parkinson's disease (PD), progressive supranuclear palsy (PSP), corticobasal dementia (CBD), multiple system atrophy (MSA) and vascular parkinsonism (VP). Each of these diseases has a singular physiopathological origin, course and prognosis. Numerous imaging studies consequently aimed at finding markers to early make the distinction between the different types of parkinsonism, in order to identify patients who could benefit from dopaminergic agonist therapy.

Excessive iron deposition in the subcortical and brainstem nuclei has been described in numerous neurodegenerative disorders including Parkinson's disease. Increased iron levels are more frequent in area that are rich in dopaminergic neurons and have been implicated in the development of movement disorders, the distribution of areas with increased iron deposition however varying according to parkinsonism types. Iron deposition quantification could thus potentially help in differentiating parkinsonism types and could improve therapy guidance. Quantitative susceptibility mapping (QSM) locally estimates the magnetic susceptibility of brain tissues based on gradient-echo signal phase. The local susceptibility being sensitive to the presence of paramagnetic susbtances, QSM allows the non-invasive evaluation of iron distribution and quantification in the brain with high image quality (Liu et al., 2013). However, since iron deposition followed an exponential curve during normal aging in most of the basal ganglia the potential of QSM to distinguish between healthy and parkinsonian subjects in elderly remains unclear.

The aim of this study was thus to determine susceptibility values in the basal ganglia of elderly patients with parkinsonian syndromes, to compare these values to healthy aged-matched controls and between parkinsonian syndrome types. Secondly, investigators aimed to evaluate microstructural changes in the basal ganglia using diffusion tensor imaging (DTI) in the same population and to determine whether susceptibility and DTI parameter changes are correlated. Finally investigators sought to assess the relation between susceptibility/DTI parameter values in the basal ganglia and behavioral measures of motor and cognitive abilities.

DETAILED DESCRIPTION:
Elderly patients with parkinsonian syndrome and healthy age-matched controls are enrolled in this study. The subjects all undergo a brain MRI exam. Controls are selected to match the age distribution of patients.

Clinical evaluation The day of the brain MRI examination, all patients undergo a neurological and neuropsychological evaluation. Diagnoses are established by a neurologist experienced with parkinsonian syndromes according to established guidelines: the UK Parkinson's Disease Society Brain Bank criteria for idiopathic PD, the National Institute of Neurological Disorders and Stroke and the Society for Progressive Supranuclear Palsy criteria for progressive supranuclear palsy, Lang's criteria for corticobasal dementia, Gilman's criteria for multiple system atrophy and Zijlmans's criteria for vascular parkinsonism.

Impairment of the motor function related to parkinsonian syndrome is assessed using the Hoehn and Yahr scale (range 0-5), the Schwab and England Activities of Daily Living scale (range 0-100%), the Unified Parkinson's Disease Rating Scale (UPDRS, range 0-199) and the Short Motor Disability scale (range 0-17).

Cognitive impairment is assessed using the Mini Mental Sate Examination (MMSE) score (range 0-30), the Grober and Buschke verbal-learning test (range 0-16), a semantic-processing task (LEXIS test, range 0-64), the forward/backward Digit span task (range 0-17) of the third Wechsler Adult Intelligence Scale and the Rey-Osterrieth Complex-Figure (ROCF) test (range 0-36) to assess visuospatial abilities, attention, executive function and working memory.

The Mattis Dementia-Rating scale (range 0-144) and the Beck Depression Inventory (range 0-63) are performed to look for depression. The Educational Attainment and the National Institute of Health Stroke Score (NIHSS) (range 0-42) are also recorded.

MRI acquisition and processing. All patients undergo a brain MRI on a 3-Tesla scanner including 3D triple echo gradient echo acquisition to generate susceptibility weighted images, T1-weighted magnetisation-prepared rapid 3D gradient-echo (MPRAGE) and diffusion tensor imaging acquisition.

Susceptibility weighted imaging raw data are preprocessed to obtain magnitude and phase images for each echo time. Quantitative susceptibility maps are then generated using SPM8 software (Statistical Parametric Mapping, Wellcome Department of Cognitive Neurology, Institute of Neurology, London, UK; http://www.fil.ion.ucl.ac.uk/spm/, Matlab 2014a, The MathWorks, Natick, MA, USA).

ELIGIBILITY:
Inclusion Criteria:

* For Both patients and healthy volunteers :

  * Age limits ≥ 70 et ≤ 90 years
  * Subject able to understand the nature, the aim and the methodology of the study.
  * Collection of the infomed consent
  * Affiliation or recipient with the mode of social security.
* For the patients :

Parkinsonian Syndrome began after 65 years defined as Parkinson's disease Multiple System Atrophy (AMS), Progressive Supranuclear Palsy, Vascular Parkinson

* For the healthy volunteers :

The healthy volunteers will be selected according to the age and the of the study's patients.

Exclusion Criteria:

* For Both patients and healthy volunteers :

  * Person with majority age protected by the law (supervision or trusteeship).
  * Loss of liberty per court order or administative
  * Subject presenting contraindications in MRI (valve of ventricular diversion, Ferromagnetic foreign bodies, pace-maker, Implantable defibrillator (ICD), Cochlear hearing implant, Claustrophobia, ….)
  * Antecedent of serious cranial trauma (according to classification) of ischeamic stroke ou intracranial hematoma.
* For the patients :

  •Patient treated by neuroleptics
* For the healthy volunteers :

  * Antecedent of neurological desease
  * Antecedent of psychiatric trouble de trouble psychiatrique (Except anxio-depressive disorder)
  * In period of exclusion relative to another protocol or which the annual amount of the allowances maximum of 4500 € was reached.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Quantitative susceptibility mapping | 1 month
  Susceptibility weighted imaging raw data are preprocessed to obtain magnitude and phase images for each echo time. Quantitative susceptibility maps are then generated using a in-house software.

SECONDARY OUTCOMES:
Diffusion tensor imaging | 1 month
  Diffusion tensor imaging data are acquired and corrected for distortions due to eddy currents in the gradient coils. They are processed using FSL software to generate fractional anisotropy (FA), mean diffusivity (MD) and the three eigenvalues (λ1, λ2, λ3) used to calculate axial diffusivity (AD=λ1) and radial diffusivity (RD=[λ2 + λ3]/2) maps.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Menjot de Champfleur, Medical PHD, Principal Investigator — UH Montpellier
Locations (1):
- Service de Neuroradiologie, Hopital Gui de Chauliac, CHU de Montpellier, Montpellier, France, France